CLINICAL TRIAL: NCT03323983
Title: Exploratory Study on Link Between Dynamic Hyperinflation and Lung Clearance Index in Cystic Fibrosis (Étude du Lien Entre la Distension Dynamique et l'Indice de Clairance Pulmonaire Dans la Mucoviscidose)
Brief Title: Exploratory Study on Link Between Dynamic Hyperinflation and Lung Clearance Index in Cystic Fibrosis
Acronym: ICP2DM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2016/293
Record Dates: First submitted 2017-10-25; First posted 2017-10-27 (Actual); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Cystic Fibrosis; Lung Clearance Index
MeSH Terms: conditions — Cystic Fibrosis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal lung clearance index
  Interventions: Other: data collection
- Elevated lung clearance index
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — data collection

SUMMARY:
Recent improvements in cystic fibrosis management have enabled an important subset of patients to maintain normal spirometry. Nevertheless, even in these patients with normal spirometry, chest computed tomography (CT) might identify structural lung abnormalities such as bronchiectasis, mucus plugging, bronchiolitis and air trapping.

Lung clearance index (LCI) has been shown to correlate well with structural pulmonary alterations seen on CT even in CF patients with well-preserved spirometry. In cystic fibrosis, a high LCI is associated with a worse feeling of illness assessed by the Cystic Fibrosis Questionnaire-Revised (CFQ-R). School-aged CF patients with normal spirometry also have normal aerobic function as assessed by peak oxygen uptake (V̇O2) measured during symptom-limited incremental cardiopulmonary exercise test. However, the ability of LCI to predict ventilatory abnormalities appearing at exercise in CF patients has not been investigated. The investigators therefore aimed to compare physiological parameters at exercise between CF patients with elevated LCI (i.e., LCI above the upper limit of normal [ULN]) and patients with normal LCI, all with preserved spirometry.

ELIGIBILITY:
Inclusion Criteria:

* children between 10 to 17 years old with a diagnosis of cystic fibrosis confirmed by sweat test and genetic test
* pulmonary function test and incremental cardiopulmonary exercise test included in their follow-up
* lung function preserved (FEV1 greater than the lower limit of normal)
* affiliation to the French social security
* children and their legal guardians informed of the use of anonymised data

Exclusion Criteria:

* recent respiratory infection
* association with another obstructive respiratory disease, especially with asthma

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children between 10 to 17 years old with a diagnosis of cystic fibrosis
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
The main objective is to explore the relationship between elevated lung clearance index and dynamic hyperinflation in cystic fibrosis patients with preserved pulmonary function. | day 1

IPD SHARING:
Plan to Share IPD: No